CLINICAL TRIAL: NCT02958020
Title: Multicenter Cohort Study on Osteoporosis in the Middle-aged and Elderly People in Shanghai, China
Brief Title: Multicenter Cohort Study on Osteoporosis
Status: Recruiting | Type: Observational
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Collaborators: Wangjing Hospital, China Academy of Chinese Medical Sciences (Other); Dongzhimen Hospital, Beijing (Other); The First Affiliated Hospital of Guangzhou University of TCM (Unknown); Guangdong Provincial Hospital of Traditional Chinese Medicine (Other); Affiliated Hospital of Changchun University of Chinese Medicine (Other); Gansu Provincial Hospital (Other); Guangzhou Kingmed Diagnostics Co., Ltd. (Unknown); Affiliated Hospital of Shandong University of Traditional Chinese Medicine (Other); Yunnan Provincial Hospital of Traditional Chinese Medicine (Unknown); Shenzhen Pingle Orthopedic Hospital (Unknown); First People's Hospital of Nankang District, Ganzhou City (Unknown)
Responsible Party: Principal Investigator, Bing Shu, Associate Professor, Shanghai University of Traditional Chinese Medicine
Other Study IDs: osteoporosis cohort
Record Dates: First submitted 2016-11-03; First posted 2016-11-08 (Estimated); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Osteoporosis
Keywords: cohort, osteoporosis, bone mineral density, Chinese
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA from blood cells will be preserved for specific study including SNP ananlyses.Tongue coating and feces will be preserved for microflora analyses.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a multicenter cohort study on osteoporosis in nine cities of China which locate in the east, south, north, west, middle of China. At least 3000 middle-aged and elderly permanent residents (women aged from 45 to 79, and men aged from 50 to 79) in every city will be enrolled. Residents with severe mental diseases, physical diseases or acute infectious diseases who could not cooperate with the survey as well as lactating or pregnant women were excluded. All the enrolled residents who signed informed consent will finish questionnaire including demographic characteristics, history of smoking, alcohol drinking, falls and fracture, family genetic history, chronic diseases and medicine,diary and physical practice，stool and urine status. Osteoporosis risk, health status, constitution of traditional Chinese medicine (TCM),symptoms of kidney yang deficiency in TCM，living environment,sweating status will be evaluated. Fasting blood glucose test and other blood tests for liver and kidney function,bone metabolism，vitamins，vitamin D metabolism and transportation as well as calcium and phosphate metabolism, will be performed. Bone mineral density and physical examinations (height, weight, waist circumference, hip circumference,grip,sit-to-stand test, tongue coating and pulse) will also be performed at enrollment and every two years after enrollment. DNA of blood cells will be preserved for specific study such as SNP analyses.Tongue coating and feces will be preserved for microflora analyses.

ELIGIBILITY:
Inclusion Criteria:

* permanent residents
* women aged from 45 to 79, and men aged from 50 to 79

Exclusion Criteria:

* severe mental diseases, physical diseases or acute infectious diseases who could not cooperate with the survey.
* lactating or pregnant women.

Ages: 45 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Nine cities which locate in the east, south, north, west and middle of China were involved. In each city, at least 3000 middle-aged and elderly permanent residents were enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2016-11 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
changes in bone mineral density from baseline to 2, 4, 6, 8 and 10 years after enrollment | at enrollment, and 2, 4, 6, 8 and 10 years after enrollment
  lumbar (L1-4 as well as total) and hip bone mineral density will be recorded by dual energy X-ray absorptiometry.

SECONDARY OUTCOMES:
fracture questionnaire | at enrollment, and 2, 4, 6, 8 and 10 years after enrollment
  information about fracture including cause, time, skeletal site and therapy during the follow-up period will be collected through fracture questionnaire
serum osteocalcin | at enrollment, and 2, 4, 6, 8 and 10 years after enrollment
serum procollagen type I N-terminal propeptide (PINP) | at enrollment, and 2, 4, 6, 8 and 10 years after enrollment
serum bone alkaline phosphatase (BALP) | at enrollment, and 2, 4, 6, 8 and 10 years after enrollment
serum β-crosslaps (β-CTX) | at enrollment, and 2, 4, 6, 8 and 10 years after enrollment
serum Ca | at enrollment, and 2, 4, 6, 8 and 10 years after enrollment
serum P | at enrollment, and 2, 4, 6, 8 and 10 years after enrollment
serum Mg | at enrollment, and 2, 4, 6, 8 and 10 years after enrollment
serum fibroblast growth factor (FGF)23 | at enrollment, and 2, 4, 6, 8 and 10 years after enrollment
serum parathormone (PTH) | at enrollment, and 2, 4, 6, 8 and 10 years after enrollment
serum total 25(OH) vitamin D | at enrollment, and 2, 4, 6, 8 and 10 years after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Yongjun Wang, Principal Investigator — Shanhgai University of TCM
Locations (12):
- China (12):
  - Shenzhen Pingle Orthopedic Hospital, Shenzhen, Guangdong
  - First People's Hospital of Nankang District, Ganzhou City, Ganzhou, Jiangxi
  - Shandong Provincial Hospital of Traditional Chinese Medicine, Jinan, Shandong
  - Yunnan Provincial Hospital of Traditional Chinese Medicine, Kunming, Yunnan
  - Dongzhimen Hospital, Beijing, Beijing
  - Wangjing Hospital, China Academy of Chinese Medical Sciences, Beijing
  - Affiliated Hospital of Changchun University of Traditional Chinese Medicine, Changchun
  - Guangdong Provincial Hospital of Traditional Chinese Medicine, Guangzhou
  - Guangzhou Kingmed Diagnostics Co., Ltd., Guangzhou
  - The First Affiliated Hospital of Guangzhou University of Traditional Chinese Medicine, Guangzhou
  - Gansu Provincial Hospital of Traditional Chinese Medicine, Lanzhou
  - Longhua Hospital, Shanghai University of TCM, Shanghai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang J, Shu B, Li CG, Xie XW, Liang D, Chen BL, Lin XC, Wei X, Wang L, Leng XY, Zhou YJ, Chen PZ, Tao YR, Zhou Y, Zhang Y, Cui XJ, Lu S, Wang H, Shi Q, Wang YJ. Polymorphisms of genes related to vitamin D metabolism and transportation and its relationship with the risk of osteoporosis: protocol for a multicentre prospective cohort study in China. BMJ Open. 2019 Nov 24;9(11):e028084. doi: 10.1136/bmjopen-2018-028084. PMID 31767578
- [Derived] Wang J, Chen L, Zhang Y, Li CG, Zhang H, Wang Q, Qi X, Qiao L, Da WW, Cui XJ, Lu S, Wang YJ, Shu B. Association between serum vitamin B6 concentration and risk of osteoporosis in the middle-aged and older people in China: a cross-sectional study. BMJ Open. 2019 Jul 4;9(7):e028129. doi: 10.1136/bmjopen-2018-028129. PMID 31278103